CLINICAL TRIAL: NCT01396720
Title: Impact of Citalopharm and Fluvoxamine on Platelet Response to Clopidogrel, a Randomized, Double-blind, Crossover Trial
Brief Title: Impact of Citalopharm and Fluvoxamine on Platelet Response to Clopidogrel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, RONNY ALCALAI, Director, Cardiac Care Unit, Mt. Scopus, Hadassah Medical Organization
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0255-HMO-CTIL
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Drug Interactions Between Clopidogrel and Serotonin Reuptake Inhibitors
MeSH Terms: interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluvoxamine (Active Comparator)
  Interventions: Drug: fluvoxamine
- citalopharm (Active Comparator)
  Interventions: Drug: citalopharm

INTERVENTIONS:
Drug: fluvoxamine — Fluvoxamine 100mg daily, 7 days
  Arms: fluvoxamine
Drug: citalopharm — Citalopharm 20mg daily, 7 days
  Arms: citalopharm

SUMMARY:
Clopidogrel is a platelets inhibitor that is widely used particularly during and after acute coronary events and coronary interventions. Several studies have shown that some patients are resistant to clopidogrel. The resistance mechanism is not entirely clear, but at least in part it is related to interactions between medications. Clopidogrel is a pro-drug converted in vivo to its active metabolite by CYP2C19 and CYP3A in the liver. Consequently drugs that inhibit the CYP2C19 can affect the production of the active metabolite and cause "clopidogrel resistance". Therefore the FDA has recently published a "safety alert" which recommends avoiding cross treatment with clopidogrel and drugs that are expected to inhibit CYP2C19 (including omeprazole, fluvoxamine, cimetidine, fluconazole and others). Nevertheless there no clear evidence in the literature for clinical relevance of such interactions.

Selective serotonin reuptake inhibitors (SSRIs) are group of antidepressant drugs that are widely used for treatment of depression and anxiety. SSRIs are considered to be very safe with favorable side effect profile, hence many patient after coronary events who suffers from behavioral and emotional disturbances are treated with those drugs. However there are several reports that SSRIs can inhibit platelet function and increase bleeding tendency particularly in concomitant administration with aspirin. The proposed mechanism is blocking of platelets serotonin reuptake that result in platelet dysfunction.

Fluvoxamine - is a member in the SSRI family and a potent inhibitor of the CYP2C19. Theoretically fluvoxamine should have two conflicting effects on the response to clopidogrel. Pharmacokinetically it is expected to decrease the clopidogrel responsiveness due to inhibition of CYP2C19 and reduction in the production of the active metabolite. On the other hand "pharmacodynamically" fluvoxamine may directly inhibit platelet aggregation due its effect on serotonin reuptake, thus increasing the effect of clopidogrel. Other SSRIs that do not interact with the CYP2C19 such as citalophram are expected to have only pharmocodynamic effect on platelet aggregation.

Although both clopidogrel and SSRIs are widely used in the last decade and concomitant treatment is quite common, no data is available about in influence of the interaction between those drugs on platelet function and on clinical events. The net effect of fluvoxamine and other SSRIs on platelet function in the presence of clopidogrel is not known.

The aim of the investigators study is to assess the effect of two SSRIs fluvoxamine and citalophram on platelet aggregation and to test the effect of these drugs on the laboratory response to clopidogrel, in healthy individuals.

Study design: randomized, double blinded, controlled crossover trial. Primary study end point: Change in % platelet aggregation and VASP phosphorylation after treatment with clopidogrel + fluvoxamine or clopidogrel + citalophram as compared to each drug alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Bleeding tendency
* Hypersensitivity to study drugs

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity in response to clopidogrel | 12 months
  We will assess response to clopidogrel by two methods: 1. % change in platelet aggregation using light transmission aggregometry with ADP as agonist. 2. % of change in VASP phosphorylation - measure of activation of the platelet P2Y12 receptor (targeted by clopidogrel). The response clopidogrel will be measured after administration of clopidogrel and after co-administration of clopidogrel and each of the study drugs (fluvoxamine and citalophram). Statistical analysis will be performed to assess differences in platelet function between the different drug treatments.

REFERENCES:
- [Derived] Hirsh-Rokach B, Spectre G, Shai E, Lotan A, Ritter A, Al-Aieshy F, Malmstrom RE, Varon D, Alcalai R. Differential impact of selective serotonin reuptake inhibitors on platelet response to clopidogrel: a randomized, double-blind, crossover trial. Pharmacotherapy. 2015 Feb;35(2):140-7. doi: 10.1002/phar.1542. PMID 25689244